CLINICAL TRIAL: NCT00696878
Title: A Phase III, Uncontrolled Trial to Assess the Non-immunogenicity and Safety of Org 36286 in Patients Undergoing Repeated Controlled Ovarian Stimulation Cycles Using a Multiple Dose GnRH Antagonist Protocol
Brief Title: Corifollitropin Alfa in Participants Undergoing Repeated Controlled Ovarian Stimulation (COS) Cycles Using a Multiple Dose Gonadatropin Releasing Hormone (GnRH) Antagonist Protocol (Study 38825)(P05714)
Acronym: Trust
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05714; MK-8962-007 (Other: Merck Study Number); 38825 (Other: Merck Study Number); 2004-004966-34 (EudraCT Number)
Record Dates: First submitted 2008-06-11; First posted 2008-06-13 (Estimated); Results first posted 2015-04-23 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2022-02

CONDITIONS: In Vitro Fertilization
Keywords: Infertility; Pharmacological effects of drugs; Hormones, Hormone Substitutes and Hormone Antagonists; Pharmacological Actions; Multi-center
MeSH Terms: conditions — Infertility | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Corifollitropin alfa 150 µg (Experimental): Up to 3 COS cycles (also called treatment cycles) were performed, each including the following: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of GnRH antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of recombinant Human Chorion Gonadotropin ([rec]hCG) (5,000-10,000 IU/250 µg). Administration of (rec)hCG occurred when 3 follicles ≥17 mm were observed on ultrasound scan (USS). Daily dosing with Follicle Stimulating Hormone (FSH) (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone for luteal phase support was administered starting on the day of oocyte pick-up (34-36 hours after [rec]hCG) and continued for approximately 6 weeks. After COS cycles 1 and 2, Frozen-Thawed Embryo Transfer cycles (up to 3 after each COS cycle) could occur.
  Interventions: Drug: Corifollitropin alfa; Biological: FSH; Biological: GnRH antagonist; Biological: (rec)hCG; Drug: Progesterone

INTERVENTIONS:
Drug: Corifollitropin alfa — Corifollitropin alfa 150 µg administered as a single subcutaneous dose.
  Other Names: Org 36286; SCH 900962; MK-8962
Biological: FSH — FSH administerd subcutaneously at a dose not to exceed 225 IU/day.
Biological: GnRH antagonist — GnRH antagonist administered subcutaneously at a dose of 0.25 mg/day.
Biological: (rec)hCG — (rec)hCG administered subcutaneously at a dose of 5,000-10,000 IU/250 µg.
Drug: Progesterone — Progesterone administered vaginally at a dose of at least 600 mg/day.

SUMMARY:
The objective of the trial is to assess the non-immunogenicity and safety of corifollitropin alfa (also known as Org 36286, SCH 900962 and MK-8962) in participants undergoing repeated COS cycles using a multiple dose GnRH antagonist protocol.

DETAILED DESCRIPTION:
This trial is designed as an open-label, uncontrolled, repeated cycle trial to assess the non-immunogenicity and safety of corifollitropin alfa in participants undergoing repeated COS cycles for in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI) using a multiple dose GnRH antagonist protocol. The trial period per participant will cover 1, 2 or 3 COS treatment cycles and no more than three (in-between two stimulation cycles) Frozen-Thawed Embryo Transfer (FTET) cycles following either or both of the first two treatment cycles. In each stimulation cycle, participants receive a single injection of corifollitropin alfa and one week later, treatment is continued with a daily dose of any FSH-containing preparation up to the day of (rec)hCG administration for final oocyte maturation. Assessment of anti-corifollitropin alfa antibodies and local tolerance after corifollitropin alfa injection are important safety endpoints in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Females of couples with an indication for COS and IVF or ICSI;
* >=18 and <=39 years of age at the time of signing informed consent;
* Body weight > 60 kg and body mass index (BMI) >=18 and <=29 kg/m^2;
* Normal menstrual cycle length: 24-35 days;
* Availability of ejaculatory sperm (use of donated and/or cryopreserved sperm is allowed);
* Willing and able to sign informed consent.

Exclusion Criteria:

* History of or any current (treated) endocrine abnormality;
* History of ovarian hyper-response or history of ovarian hyperstimulation syndrome (OHSS);
* History of or current polycystic ovary syndrome (PCOS);
* More than 20 basal antral follicles (size: <11 mm, both ovaries combined) as measured on USS in the early follicular phase (menstrual cycle day 2-5);
* Less than 2 ovaries or any other ovarian abnormality, including endometrioma >10 mm (visible on USS);
* Presence of unilateral or bilateral hydrosalpinx (visible on USS);
* More than three unsuccessful COS cycles since the last established ongoing pregnancy (if applicable);
* History of non- or low ovarian response to FSH/human menopausal gonadotrophin (hMG) treatment;
* FSH > 12 IU/L or luteinizing hormone (LH) > 12 IU/L as measured by the local laboratory (sample taken during the early follicular phase: menstrual cycle day 2-5);
* Any clinically relevant abnormal laboratory value based on a sample taken during the screening phase, including abnormal cervical smear (Papanicolaou [PAP]>=III, cervical intraepithelial neoplasia [CIN]>=1);
* Contraindications for the use of gonadotropins (e.g. tumors, pregnancy/lactation, undiagnosed vaginal bleeding, hypersensitivity, ovarian cysts) or GnRH antagonists (e.g. hypersensitivity, pregnancy/lactation);
* Recent history of or current epilepsy, human immunodeficiency virus (HIV) infection, thrombophilia, diabetes or cardiovascular, gastro-intestinal, hepatic, renal, or pulmonary disease;
* Abnormal karyotyping of the participant or her partner (if karyotyping is performed);
* History or presence of alcohol or drug abuse within 12 months prior to signing informed consent;
* Previous use of corifollitropin alfa;
* Use of hormonal preparations within 1 month prior to screening;
* Administration of investigational drugs within three months prior to signing informed consent.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 682 (Actual)
Dates: Start 2006-09-26 (Actual); Primary Completion 2009-02-17 (Actual); Study Completion 2009-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zandvliet AS, Prohn M, de Greef R, van Aarle F, McCrary Sisk C, Stegmann BJ. Impact of patient characteristics on the pharmacokinetics of corifollitropin alfa during controlled ovarian stimulation. Br J Clin Pharmacol. 2016 Jul;82(1):74-82. doi: 10.1111/bcp.12939. Epub 2016 May 31. PMID 26991902
- [Derived] Griesinger G, Verweij PJ, Gates D, Devroey P, Gordon K, Stegmann BJ, Tarlatzis BC. Prediction of Ovarian Hyperstimulation Syndrome in Patients Treated with Corifollitropin alfa or rFSH in a GnRH Antagonist Protocol. PLoS One. 2016 Mar 7;11(3):e0149615. doi: 10.1371/journal.pone.0149615. eCollection 2016. PMID 26950065
- [Derived] Rombauts L, Lambalk CB, Schultze-Mosgau A, van Kuijk J, Verweij P, Gates D, Gordon K, Griesinger G. Intercycle variability of the ovarian response in patients undergoing repeated stimulation with corifollitropin alfa in a gonadotropin-releasing hormone antagonist protocol. Fertil Steril. 2015 Oct;104(4):884-890.e2. doi: 10.1016/j.fertnstert.2015.06.027. Epub 2015 Jul 15. PMID 26187300
- [Derived] Norman RJ, Zegers-Hochschild F, Salle BS, Elbers J, Heijnen E, Marintcheva-Petrova M, Mannaerts B; Trust Investigators. Repeated ovarian stimulation with corifollitropin alfa in patients in a GnRH antagonist protocol: no concern for immunogenicity. Hum Reprod. 2011 Aug;26(8):2200-8. doi: 10.1093/humrep/der163. Epub 2011 May 27. PMID 21622693

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: To complete study, a participant must have embryo transfer in the 3rd Controlled Ovarian Stimulation (COS) cycle (Treatment Cycle 3).
Groups:
- Corifollitropin Alfa 150 µg: Up to 3 COS cycles (also called treatment cycles) were performed, each including the following: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of Gonadotropin Releasing Hormone (GnRH) antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of recombinant Human Chorion Gonadotropin ([rec]hCG) (5,000-10,000 IU/250 µg). Daily dosing with Follicle Stimulating Hormone (FSH) (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone was administered for luteal phase support. After COS cycles 1 and 2, Frozen-Thawed Embryo Transfer (FTET) cycles (up to 3 after each COS cycle) could occur.
Period: Overall Study
Arm/Group | Corifollitropin Alfa 150 µg
Started | 682
Completed | 178
Not Completed | 504
Not completed — Adverse Event | 8
Not completed — Withdrawal by Subject | 87
Not completed — Stop Treat Cycle 3 not for Adverse Event | 18
Not completed — Pregnant prior to Treat Cycle 3 | 304
Not completed — Trial stopped | 32
Not completed — Other reason (not specified) | 55

BASELINE CHARACTERISTICS:
Groups:
- Corifollitropin Alfa 150 µg: Up to 3 COS cycles (also called treatment cycles) were performed, each including the following: A single injection of 150 µg corifollitropin alfa was administered on Day 2 or 3 of the menstrual cycle (Stimulation Day 1). Administration of GnRH antagonist (0.25 mg/day) started on Stimulation Day 5 or 6 and continued through day of administration of (rec)hCG (5,000-10,000 IU/250 µg). Daily dosing with FSH (not to exceed 225 IU/day) began on Stimulation Day 8 and continued up to day of (rec)hCG administration. Progesterone was administered for luteal phase support. After COS cycles 1 and 2, FTET cycles (up to 3 after each COS cycle) could occur.
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.9 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 682
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinically Relevant Immunogenicity
Description: Serum samples obtained pre-dose and at 2 weeks after embryo transfer (ET), or at cycle discontinuation and 2-3 weeks after cycle discontinuation if cycle was stopped before ET was performed, were analyzed for presence of anti-corifollitropin alfa antibodies using screening and confirmatory tests. If a participant was confirmed to have anti-corifollitropin alfa antibody present in a post dose sample according to these tests, review of adverse events (AEs) in the participant was performed. The sample was also tested to evaluate whether the antibody appeared to have neutralizing activity that would interfere with the study drug biological effect. A participant was determined to have clinically relevant immunogenicity if the participant had a confirmed post dose anti-corifollitropin alfa antibody test result accompanied by clinical signs of immunogenicity (e.g., hypersensitivity reaction), considering also the results of the test for neutralizing activity of any antibody present.
Time Frame: Pre-dose (Stimulation Day 1) and up to approximately 40 days post dose in each treatment cycle
Population: Participants who received corifollitropin alfa and had a post dose sample for anti-corifollitropin alfa antibody testing
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
percentage of participants
  Cycle 1 (n=681) | 0.0
  Cycle 2 (n=372) | 0.0
  Cycle 3 (n=192) | 0.0
Statistical Analysis 1: Comparison: Corifollitropin Alfa 150 µg; During sample size determination, the upper limit of the one-sided 95% confidence interval for the population incidence of immunogenicity, if no immunogenicity is observed, was calculated. If no immunogenicity is observed in the projected 150 participants who receive corifollitropin alfa during 3 COS cycles, then the upper limit for the population is 2%. For the projected 300 participants who receive corifollitropin alfa during 2 COS cycles, the upper limit for the population is 1%; Test type: Superiority or Other; Percentage with immunogenicity = 0.0, 95% CI 1-sided [upper limit 0.4] — Provided limit is upper 1-sided 95% confidence limit for study population for percentage of participants with clinically relevant immunogenicity, after Cycle 1
Statistical Analysis 2: Comparison: Corifollitropin Alfa 150 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percentage with immunogenicity = 0.0, 95% CI 1-sided [upper limit 0.8] — Provided limit is upper 1-sided 95% confidence limit for study population for percentage of participants with clinically relevant immunogenicity, after Cycle 2
Statistical Analysis 3: Comparison: Corifollitropin Alfa 150 µg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Percentage with immunogenicity = 0.0, 95% CI 1-sided [upper limit 1.5] — Provided limit is upper 1-sided 95% confidence limit for study population for percentage of participants with clinically relevant immunogenicity, after Cycle 3

2. Primary Outcome: Local Tolerance at Injection Site: Number of Participants With no Event of Itching and With Mild, Moderate and Severe Itching in Any of 3 Treatment Cycles
Description: At 30 minutes after dosing in each treatment cycle, the corifollitropin alfa injection site was assessed for the presence of itching, pain, redness and swelling, each of which was scored as none (no event), mild, moderate or severe. This measure reports results for the assessment of itching. A participant with an event was counted once in this analysis.
Time Frame: 30 minutes post dose in each treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  None | 679
  Mild | 3
  Moderate | 0
  Severe | 0

3. Primary Outcome: Local Tolerance at Injection Site: Number of Participants With no Event of Pain and With Mild, Moderate and Severe Pain in Any of 3 Treatment Cycles
Description: At 30 minutes after dosing in each treatment cycle, the corifollitropin alfa injection site was assessed for the presence of itching, pain, redness and swelling, each of which was scored as none (no event), mild, moderate or severe. This measure reports results for the assessment of pain. A participant with an event was counted once in this analysis.
Time Frame: 30 minutes post dose in each treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  None | 678
  Mild | 4
  Moderate | 0
  Severe | 0

4. Primary Outcome: Local Tolerance at Injection Site: Number of Participants With no Event of Redness and With Mild, Moderate and Severe Redness in Any of 3 Treatment Cycles
Description: At 30 minutes after dosing in each treatment cycle, the corifollitropin alfa injection site was assessed for the presence of itching, pain, redness and swelling, each of which was scored as none (no event), mild, moderate or severe. This measure reports results for the assessment of redness. A participant with an event was counted once in this analysis.
Time Frame: 30 minutes post dose in each treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  None | 654
  Mild | 28
  Moderate | 0
  Severe | 0

5. Primary Outcome: Local Tolerance at Injection Site: Number of Participants With no Event of Swelling and With Mild, Moderate and Severe Swelling in Any of 3 Treatment Cycles
Description: At 30 minutes after dosing in each treatment cycle, the corifollitropin alfa injection site was assessed for the presence of itching, pain, redness and swelling, each of which was scored as none (no event), mild, moderate or severe. This measure reports results for the assessment of swelling. A participant with an event was counted once in this analysis.
Time Frame: 30 minutes post dose in each treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  None | 680
  Mild | 2
  Moderate | 0
  Severe | 0

6. Primary Outcome: Local Tolerance at Injection Site Overall Summary: Number of Participants With no Local Tolerance Event (Itching, Pain, Redness or Swelling) and With a Mild, Moderate and Severe Local Tolerance Event in Any of 3 Treatment Cycles
Description: At 30 minutes after dosing in each treatment cycle, the corifollitropin alfa injection site was assessed for the presence of itching, pain, redness and swelling, each of which was scored as none (no event), mild, moderate or severe. This measure reports results considering the occurrence of any of the defined local tolerance events. A participant with an event was counted once in this analysis.
Time Frame: 30 minutes post dose in each treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  None | 647
  Mild | 35
  Moderate | 0
  Severe | 0

7. Primary Outcome: Number of Participants With AEs
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: Up to approximately 26 months after first dose of corifollitropin alfa
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants | 409

8. Primary Outcome: Number of Participants With Serious AEs (SAEs)
Description: An SAE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, or was a congenital anomaly/birth defect. SAEs that occurred in fetuses or infants during the study period are included in this summary of SAEs, and are allocated to the associated study participant who was administered corifollitropin alfa.
Time Frame: Up to approximately 26 months after first dose of corifollitropin alfa
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants | 51

9. Primary Outcome: Number of Participants With Moderate to Severe Ovarian Hyperstimulation Syndrome (OHSS)
Description: OHSS was classified on study based on a slightly modified WHO Scientific Group (1973) classification: Grade I (mild) = characterized by excessive steroid secretion and ovarian enlargement (5-7 cm). Abdominal discomfort, including abdominal pain, is present. Grade II (moderate) = characterized by distinct ovarian cysts (ovary size 8-10 cm), accompanied by abdominal pain and tension, nausea, vomiting, diarrhea. Grade III (severe) = characterized by enlarged cystic ovaries (ovary size >10 cm), accompanied by ascites and occasionally hydrothorax. Abdominal tension and pain may be severe. Pronounced hydrothorax together with an abdominal cavity filled with cysts and fluid elevating the diaphragm may cause severe breathing difficulties. Large quantities of fluid inside the cysts and in the peritoneal and pleural cavities cause haemoconcentration and increased blood viscosity. In rare cases, the syndrome may further be complicated by the occurrence of thromboembolic phenomena.
Time Frame: Up to approximately 1 month after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), within a treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  Cycle 1 (n=682) | 12
  Cycle 2 (n=375) | 4
  Cycle 3 (n=198) | 0

10. Secondary Outcome: Amount of (Rec)FSH Needed From Stimulation Day 8 Onwards to Reach the Criterion for Administration of (Rec)hCG
Description: Beginning on Stimulation Day 8 of each treatment cycle, (rec)FSH was administered daily until the criteria for administration of (rec)hCG (presence of 3 follicles ≥17 mm documented by ultrasonography) was reached. The total amount of (rec)FSH administered in each participant to reach the criteria for (rec)hCG administration was calculated.
Time Frame: Stimulation Day 8 to day of (rec)hCG administration (approximately Stimulation Day 10), within a treatment cycle
Population: Participants who received corifollitropin alfa and (rec)hCG
Measure: Median (Full Range); unit: International Unit (IU)
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 664
International Unit (IU)
  Cycle 1 (n=658) | 400.0 [0 to 2100]
  Cycle 2 (n=364) | 450.0 [0 to 1950]
  Cycle 3 (n=190) | 450.0 [0 to 2250]

11. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 1 During Treatment Cycle 1
Description: For each participant, the number of follicles ≥11 mm, ≥15 mm and ≥17 mm documented by ultrasonography on defined days during the treatment cycle was calculated.
Time Frame: Stimulation Day 1 in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 1 in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 666
follicles
  follicles ≥11 mm | 0.0 (0.1)
  follicles ≥15 mm | 0.0 (0.1)
  follicles ≥17 mm | 0.0 (0.1)

12. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 1 During Treatment Cycle 2
Description: as for outcome 11
Time Frame: Stimulation Day 1 in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 1 in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 370
follicles
  follicles ≥11 mm | 0.0 (0.3)
  follicles ≥15 mm | 0.0 (0.0)
  follicles ≥17 mm | 0.0 (0.0)

13. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 1 During Treatment Cycle 3
Description: as for outcome 11
Time Frame: Stimulation Day 1 in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 1 in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 196
follicles
  follicles ≥11 mm | 0.0 (0.2)
  follicles ≥15 mm | 0.0 (0.0)
  follicles ≥17 mm | 0.0 (0.0)

14. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 5 or 6 During Treatment Cycle 1
Description: as for outcome 11
Time Frame: Stimulation Day 5 or 6 in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 5 or 6 in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 677
follicles
  follicles ≥11 mm | 5.1 (4.2)
  follicles ≥15 mm | 0.4 (1.0)
  follicles ≥17 mm | 0.1 (0.3)

15. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 5 or 6 During Treatment Cycle 2
Description: as for outcome 11
Time Frame: Stimulation Day 5 or 6 in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 5 or 6 in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 372
follicles
  follicles ≥11 mm | 4.8 (4.1)
  follicles ≥15 mm | 0.4 (1.0)
  follicles ≥17 mm | 0.1 (0.4)

16. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 5 or 6 During Treatment Cycle 3
Description: as for outcome 11
Time Frame: Stimulation Day 5 or 6 in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 5 or 6 in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 198
follicles
  follicles ≥11 mm | 4.0 (3.3)
  follicles ≥15 mm | 0.3 (0.9)
  follicles ≥17 mm | 0.0 (0.3)

17. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 8 During Treatment Cycle 1
Description: as for outcome 11
Time Frame: Stimulation Day 8 in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 8 in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 660
follicles
  follicles ≥11 mm | 11.1 (5.9)
  follicles ≥15 mm | 3.7 (3.3)
  follicles ≥17 mm | 1.1 (1.8)

18. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 8 During Treatment Cycle 2
Description: as for outcome 11
Time Frame: Stimulation Day 8 in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 8 in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 363
follicles
  follicles ≥11 mm | 10.7 (5.4)
  follicles ≥15 mm | 3.6 (3.3)
  follicles ≥17 mm | 1.2 (1.8)

19. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Stimulation Day 8 During Treatment Cycle 3
Description: as for outcome 11
Time Frame: Stimulation Day 8 in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and had data for assessment of follicles ≥11 mm on Stimulation Day 8 in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 194
follicles
  follicles ≥11 mm | 10.0 (5.8)
  follicles ≥15 mm | 3.4 (3.3)
  follicles ≥17 mm | 1.1 (1.8)

20. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Day of (Rec)hCG Administration During Treatment Cycle 1
Description: For each participant, the number of follicles ≥11 mm, ≥15 mm and ≥17 mm documented by ultrasonography on the day of (rec)hCG administration during the treatment cycle was recorded.
Time Frame: Day of (rec)hCG administration (approximately Stimulation Day 10) in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and (rec)hCG, and had data for assessment of follicles ≥11 mm on day of (rec)hCG administration in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 640
follicles
  follicles ≥11 mm | 14.5 (6.4)
  follicles ≥15 mm | 9.2 (4.3)
  follicles ≥17 mm | 5.4 (2.8)

21. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Day of (Rec)hCG Administration During Treatment Cycle 2
Description: as for outcome 20
Time Frame: Day of (rec)hCG administration (approximately Stimulation Day 10) in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and (rec)hCG, and had data for assessment of follicles ≥11 mm on day of (rec)hCG administration in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 359
follicles
  follicles ≥11 mm | 13.9 (6.0)
  follicles ≥15 mm | 9.0 (3.9)
  follicles ≥17 mm | 5.4 (2.7)

22. Secondary Outcome: Number of Follicles ≥11 mm, ≥15 mm and ≥17 mm Documented by Ultrasonography Performed in the Participant on Day of (Rec)hCG Administration During Treatment Cycle 3
Description: as for outcome 20
Time Frame: Day of (rec)hCG administration (approximately Stimulation Day 10) in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and (rec)hCG, and had data for assessment of follicles ≥11 mm on day of (rec)hCG administration in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 185
follicles
  follicles ≥11 mm | 13.7 (6.4)
  follicles ≥15 mm | 9.0 (4.7)
  follicles ≥17 mm | 5.4 (2.9)

23. Secondary Outcome: Number of Oocytes Retrieved in a Participant Among Entire Study Population
Description: Oocyte retrieval, also known as oocyte pick-up, is a technique used in in vitro fertilization (IVF) and intracytoplasmic sperm injection (ICSI) in order to remove oocytes from the ovary of the female, enabling fertilization outside the body. The number of oocytes retrieved, per participant, is summarized.
Time Frame: Day of oocyte pick-up, 34-36 hours after (rec)hCG administration (approximately Stimulation Day 10), within a treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
number of oocytes
  Cycle 1 (n=682) | 11.9 (7.2)
  Cycle 2 (n=375) | 11.5 (6.8)
  Cycle 3 (n=198) | 11.3 (7.6)

24. Secondary Outcome: Quality of Oocytes Assessed Prior to Planned ICSI in Treatment Cycle 1
Description: This measure summarizes results of assessment of the quality of oocytes performed following oocyte retrieval, among participants scheduled for ICSI in Treatment Cycle 1. For oocytes obtained from each participant, the number in each of 3 stages of oocyte development were determined. The earliest phase is the germinal vesicles stage, during which the immature oocyte appears as a large vesicular nucleus. Metaphase I is an intermediate stage during which the vesicles have broken down and the polar body has not yet formed; the oocyte is still immature. Metaphase II is the mature oocyte and is indicated by the presence of the polar body. Rating of quality for usefulness in ICSI follows the order metaphase II (best quality), metaphase I (lesser quality) and germinal vesicles stage (poorest quality). Only metaphase II oocytes can be fertilized. Metaphase I oocytes can develop in vitro to metaphase II oocytes. Germinal vesicles stage oocytes are the least useful for ICSI procedures.
Time Frame: Day of oocyte pick-up, 34-36 hours after (rec)hCG administration (approximately Stimulation Day 10), in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and were to have ICSI in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 462
number of oocytes
  Oocytes assessed | 12.2 (7.0)
  Metaphase I | 0.8 (1.4)
  Metaphase II | 9.8 (6.0)
  Germinal vesicles stage | 0.9 (1.4)

25. Secondary Outcome: Quality of Oocytes Assessed Prior to Planned ICSI in Treatment Cycle 2
Description: This measure summarizes results of assessment of the quality of oocytes performed following oocyte retrieval, among participants scheduled for ICSI in Treatment Cycle 2. For oocytes obtained from each participant, the number in each of 3 stages of oocyte development were determined. The earliest phase is the germinal vesicles stage, during which the immature oocyte appears as a large vesicular nucleus. Metaphase I is an intermediate stage during which the vesicles have broken down and the polar body has not yet formed; the oocyte is still immature. Metaphase II is the mature oocyte and is indicated by the presence of the polar body. Rating of quality for usefulness in ICSI follows the order metaphase II (best quality), metaphase I (lesser quality) and germinal vesicles stage (poorest quality). Only metaphase II oocytes can be fertilized. Metaphase I oocytes can develop in vitro to metaphase II oocytes. Germinal vesicles stage oocytes are the least useful for ICSI procedures.
Time Frame: Day of oocyte pick-up, 34-36 hours after (rec)hCG administration (approximately Stimulation Day 10), in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and were to have ICSI in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 281
number of oocytes
  Oocytes assessed | 11.6 (6.5)
  Metaphase I | 0.9 (1.5)
  Metaphase II | 9.3 (5.4)
  Germinal vesicles stage | 0.8 (1.4)

26. Secondary Outcome: Quality of Oocytes Assessed Prior to Planned ICSI in Treatment Cycle 3
Description: This measure summarizes results of assessment of the quality of oocytes performed following oocyte retrieval, among participants scheduled for ICSI in Treatment Cycle 3. For oocytes obtained from each participant, the number in each of 3 stages of oocyte development were determined. The earliest phase is the germinal vesicles stage, during which the immature oocyte appears as a large vesicular nucleus. Metaphase I is an intermediate stage during which the vesicles have broken down and the polar body has not yet formed; the oocyte is still immature. Metaphase II is the mature oocyte and is indicated by the presence of the polar body. Rating of quality for usefulness in ICSI follows the order metaphase II (best quality), metaphase I (lesser quality) and germinal vesicles stage (poorest quality). Only metaphase II oocytes can be fertilized. Metaphase I oocytes can develop in vitro to metaphase II oocytes. Germinal vesicles stage oocytes are the least useful for ICSI procedures.
Time Frame: Day of oocyte pick-up, 34-36 hours after (rec)hCG administration (approximately Stimulation Day 10), in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and were to have ICSI in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: number of oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 151
number of oocytes
  Oocytes assessed | 11.3 (6.3)
  Metaphase I | 0.8 (1.3)
  Metaphase II | 9.1 (5.2)
  Germinal vesicles stage | 0.9 (1.5)

27. Secondary Outcome: Number of Fertilized Oocytes Obtained in Treatment Cycle 1
Description: This measure presents the number of fertilized oocytes obtained per participant from the IVF or ISCI procedure, by category of number of pronuclei (PN) present: 0 PN, 1 PN, 2 PN, ≥3 PN, other (fertilized oocyte that was not placed in PN category). Normal fertilized ooctyes have 2 pronuclei (2 PN).
Time Frame: 16-18 hours after start of IVF or ICSI, which occurs on day of oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 649
number of fertilized oocytes
  0 PN fertilized oocytes | 2.2 (2.9)
  1 PN fertilized oocytes | 0.2 (0.6)
  2 PN fertilized oocytes | 6.1 (4.0)
  ≥3 PN fertilized oocytes | 0.3 (0.7)
  Other fertilized oocytes | 0.7 (1.6)

28. Secondary Outcome: Number of Fertilized Oocytes Obtained in Treatment Cycle 2
Description: This measure presents the number of fertilized oocytes obtained per participant from the IVF or ISCI procedure, by category of number of PN present: 0 PN, 1 PN, 2 PN, ≥3 PN, other (fertilized oocyte that was not placed in PN category). Normal fertilized ooctyes have 2 pronuclei (2 PN).
Time Frame: 16-18 hours after start of IVF or ICSI, which occurs on day of oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 359
number of fertilized oocytes
  0 PN fertilized oocytes | 2.1 (2.5)
  1 PN fertilized oocytes | 0.3 (0.9)
  2 PN fertilized oocytes | 6.1 (4.0)
  ≥3 PN fertilized oocytes | 0.3 (0.7)
  Other fertilized oocytes | 0.6 (1.2)

29. Secondary Outcome: Number of Fertilized Oocytes Obtained in Treatment Cycle 3
Description: as for outcome 28
Time Frame: 16-18 hours after start of IVF or ICSI, which occurs on day of oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 188
number of fertilized oocytes
  0 PN fertilized oocytes | 1.8 (2.3)
  1 PN fertilized oocytes | 0.2 (0.5)
  2 PN fertilized oocytes | 6.2 (4.2)
  ≥3 PN fertilized oocytes | 0.3 (0.7)
  Other fertilized oocytes | 0.8 (1.6)

30. Secondary Outcome: Number of Fertilized Oocytes Obtained That Were Frozen in Treatment Cycle 1
Description: This measure presents the number of fertilized oocytes obtained per participant from the IVF or ICSI procedure that were cryopreserved (frozen) for possible later use, by category of number of PN present: 0 PN, 1 PN, 2 PN, ≥3 PN, other (fertilized oocyte that was not placed in PN category). Normal fertilized ooctyes have 2 pronuclei (2 PN).
Time Frame: as for outcome 27
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 1, and were enrolled at a site using cyropreservation at the fertilized oocyte level
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 103
number of fertilized oocytes
  0 PN fertilized oocytes | 0.0 (0.0)
  1 PN fertilized oocytes | 0.0 (0.1)
  2 PN fertilized oocytes | 1.9 (3.2)
  ≥3 PN fertilized oocytes | 0.0 (0.0)
  Other fertilized oocytes | 0.0 (0.0)

31. Secondary Outcome: Number of Fertilized Oocytes Obtained That Were Frozen in Treatment Cycle 2
Description: as for outcome 30
Time Frame: as for outcome 28
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 2, and were enrolled at a site using cyropreservation at the fertilized oocyte level
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 55
number of fertilized oocytes
  0 PN fertilized oocytes | 0.0 (0.0)
  1 PN fertilized oocytes | 0.0 (0.0)
  2 PN fertilized oocytes | 1.6 (3.3)
  ≥3 PN fertilized oocytes | 0.0 (0.0)
  Other fertilized oocytes | 0.0 (0.0)

32. Secondary Outcome: Number of Fertilized Oocytes Obtained That Were Frozen in Treatment Cycle 3
Description: as for outcome 30
Time Frame: as for outcome 29
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 3, and were enrolled at a site using cyropreservation at the fertilized oocyte level
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 32
number of fertilized oocytes
  0 PN fertilized oocytes | 0.0 (0.0)
  1 PN fertilized oocytes | 0.0 (0.0)
  2 PN fertilized oocytes | 1.1 (2.1)
  ≥3 PN fertilized oocytes | 0.0 (0.0)
  Other fertilized oocytes | 0.0 (0.0)

33. Secondary Outcome: Number of Fertilized Oocytes Obtained That Were Used for Embryo Development in Treatment Cycle 1
Description: This measure presents the number of fertilized oocytes obtained per participant from the IVF or ISCI procedure that were used for embryo development, by category of number of PN present: 0 PN, 1 PN, 2 PN, ≥3 PN, other (fertilized oocyte that was not placed in PN category). Normal fertilized ooctyes have 2 pronuclei (2 PN).
Time Frame: as for outcome 27
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 649
number of fertilized oocytes
  0 PN fertilized oocytes | 0.6 (1.9)
  1 PN fertilized oocytes | 0.1 (0.3)
  2 PN fertilized oocytes | 5.7 (4.1)
  ≥3 PN fertilized oocytes | 0.0 (0.0)
  Other fertilized oocytes | 0.0 (0.1)

34. Secondary Outcome: Number of Fertilized Oocytes Obtained That Were Used for Embryo Development in Treatment Cycle 2
Description: as for outcome 33
Time Frame: as for outcome 28
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 359
number of fertilized oocytes
  0 PN fertilized oocytes | 0.6 (1.8)
  1 PN fertilized oocytes | 0.1 (0.8)
  2 PN fertilized oocytes | 5.8 (3.9)
  ≥3 PN fertilized oocytes | 0.0 (0.0)
  Other fertilized oocytes | 0.0 (0.2)

35. Secondary Outcome: Number of Fertilized Oocytes Obtained That Were Used for Embryo Development in Treatment Cycle 3
Description: as for outcome 33
Time Frame: as for outcome 29
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: number of fertilized oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 188
number of fertilized oocytes
  0 PN fertilized oocytes | 0.5 (1.6)
  1 PN fertilized oocytes | 0.1 (0.4)
  2 PN fertilized oocytes | 6.0 (4.2)
  ≥3 PN fertilized oocytes | 0.0 (0.1)
  Other fertilized oocytes | 0.1 (0.6)

36. Secondary Outcome: Fertilization Rate
Description: The fertilization rate (in percent) is defined as 100 times the ratio of the number of fertilized 2 PN oocytes obtained and the number of oocytes that was used for fertilization, per participant.
Time Frame: 16-18 hours after start of IVF or ICSI, which occurs on day of oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), within a treatment cycle
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI
Measure: Mean (Standard Deviation); unit: percentage of oocytes
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 659
percentage of oocytes
  Cycle 1 (n=649) | 67.0 (26.6)
  Cycle 2 (n=359) | 66.0 (25.8)
  Cycle 3 (n=188) | 67.3 (23.4)

37. Secondary Outcome: Number and Quality of Embryos Obtained at Day 3 After Oocyte Pick-up in Treatment Cycle 1
Description: At Day 3 after oocyte pick-up, embryos obtained from IVF or ISCI process for each participant were counted and quality was assessed. Quality was rated as Grade 1, 2 or 3, or "other grade", with Grade 1 representing the best quality. The 2 highest quality grades (Grade 1 + 2) were combined into a summary category of "good quality."
Time Frame: Day 3 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 1 and had embryo assessment at Day 3 after oocyte pick-up; excludes participants with embryo transfer or embryos cryopreserved before Day 3
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 610
number of embryos
  Total obtained | 6.4 (4.5)
  Good quality (Grade 1 + 2) | 3.2 (3.1)
  Grade 1 | 1.2 (2.1)
  Grade 2 | 1.9 (2.3)
  Grade 3 | 2.3 (2.5)
  Other grade | 1.0 (2.1)

38. Secondary Outcome: Number and Quality of Embryos Obtained at Day 3 After Oocyte Pick-up in Treatment Cycle 2
Description: as for outcome 37
Time Frame: Day 3 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 2 and had embryo assessment at Day 3 after oocyte pick-up; excludes participants with embryo transfer or embryos cryopreserved before Day 3
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 351
number of embryos
  Total obtained | 6.5 (4.4)
  Good quality (Grade 1 + 2) | 2.9 (2.8)
  Grade 1 | 1.2 (1.9)
  Grade 2 | 1.8 (2.0)
  Grade 3 | 2.4 (2.7)
  Other grade | 1.2 (2.4)

39. Secondary Outcome: Number and Quality of Embryos Obtained at Day 3 After Oocyte Pick-up in Treatment Cycle 3
Description: as for outcome 37
Time Frame: Day 3 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and had IVF and/or ICSI in Treatment Cycle 3 and had embryo assessment at Day 3 after oocyte pick-up; excludes participants with embryo transfer or embryos cryopreserved before Day 3
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 186
number of embryos
  Total obtained | 6.6 (4.8)
  Good quality (Grade 1 + 2) | 2.8 (2.7)
  Grade 1 | 1.0 (1.9)
  Grade 2 | 1.8 (2.0)
  Grade 3 | 2.6 (3.0)
  Other grade | 1.1 (2.2)

40. Secondary Outcome: Number of Embryos Transferred
Description: ET is the procedure in which one or more embryos are placed in the uterus. The number of embryos transferred, per participant, is summarized.
Time Frame: At ET, Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), within a treatment cycle
Population: Participants who received corifollitropin alfa and had ET
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 642
number of embryos
  Cycle 1 (n=616) | 1.9 (0.7)
  Cycle 2 (n=340) | 2.1 (0.7)
  Cycle 3 (n=178) | 2.2 (0.7)

41. Secondary Outcome: Number of Participants by Category of Number of Good Quality Embryos Transferred in Treatment Cycle 1
Description: The number of embryos transferred, for each participant, by category of number of "good quality" embryos transferred, is summarized. Quality was rated as Grade 1, 2 or 3, or "other grade", with Grade 1 representing the best quality. The 2 highest quality grades (Grade 1 + 2) were combined into a summary category of "good quality."
Time Frame: At ET, Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and had ET in Treatment Cycle 1
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 616
participants
  With 0 good quality embryos transferred | 110 (4.5)
  With 1 good quality embryo transferred | 230 (3.1)
  With 2 good quality embryos transferred | 201 (2.1)
  With 3 good quality embryos transferred | 75 (2.3)

42. Secondary Outcome: Number of Participants by Category of Number of Good Quality Embryos Transferred in Treatment Cycle 2
Description: as for outcome 41
Time Frame: At ET, Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and had ET in Treatment Cycle 2
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 340
participants
  With 0 good quality embryos transferred | 81 (4.5)
  With 1 good quality embryo transferred | 80 (3.1)
  With 2 good quality embryos transferred | 122 (2.1)
  With 3 good quality embryos transferred | 57 (2.3)

43. Secondary Outcome: Number of Participants by Category of Number of Good Quality Embryos Transferred in Treatment Cycle 3
Description: as for outcome 41
Time Frame: At ET, Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and had ET in Treatment Cycle 3
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 178
participants
  With 0 good quality embryos transferred | 31 (4.5)
  With 1 good quality embryo transferred | 49 (3.1)
  With 2 good quality embryos transferred | 65 (2.1)
  With 3 good quality embryos transferred | 33 (2.3)

44. Secondary Outcome: Number and Quality of Embryos Obtained That Were Frozen in Treatment Cycle 1
Description: The number of embryos that were cryopreserved (frozen) for possible later use, for each participant, overall and by embryo quality categories, is summarized. Quality was rated as Grade 1, 2 or 3, or "other grade", with Grade 1 representing the best quality. The 2 highest quality grades (Grade 1 + 2) were combined into a summary category of "good quality."
Time Frame: Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 1
Population: Participants who received corifollitropin alfa in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
number of embryos
  Total frozen | 1.6 (2.7)
  Good quality (Grade 1 + 2) | 1.2 (2.3)
  Grade 1 | 0.4 (1.2)
  Grade 2 | 0.8 (1.7)
  Grade 3 | 0.4 (1.0)
  Other grade | 0.1 (0.4)

45. Secondary Outcome: Number and Quality of Embryos Obtained That Were Frozen in Treatment Cycle 2
Description: as for outcome 44
Time Frame: Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 2
Population: Participants who received corifollitropin alfa in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 375
number of embryos
  Total frozen | 1.1 (2.1)
  Good quality (Grade 1 + 2) | 0.8 (1.7)
  Grade 1 | 0.3 (1.0)
  Grade 2 | 0.5 (1.3)
  Grade 3 | 0.3 (0.9)
  Other grade | 0.0 (0.4)

46. Secondary Outcome: Number and Quality of Embryos Obtained That Were Frozen in Treatment Cycle 3
Description: as for outcome 44
Time Frame: Day 3 or Day 5 after oocyte pick-up (34-36 hours after [rec]hCG administration [approximately Stimulation Day 10]), in Treatment Cycle 3
Population: Participants who received corifollitropin alfa in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: number of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 198
number of embryos
  Total frozen | 1.1 (2.2)
  Good quality (Grade 1 + 2) | 0.8 (1.7)
  Grade 1 | 0.3 (1.1)
  Grade 2 | 0.5 (1.3)
  Grade 3 | 0.3 (1.0)
  Other grade | 0.0 (0.4)

47. Secondary Outcome: Implantation Rate for Participants With ET
Description: The implantation rate (in percent) is defined as 100 times the maximum number of gestational sacs as assessed by any ultrasound scan after ET divided by the number of embryos transferred per participant.
Time Frame: Approximately 5-6 weeks after ET, within a treatment cycle
Population: Participants who received corifollitropin alfa and had ET
Measure: Mean (Standard Deviation); unit: percentage of embryos
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 642
percentage of embryos
  Cycle 1 (n=616) | 21.2 (36.2)
  Cycle 2 (n=340) | 16.6 (31.0)
  Cycle 3 (n=178) | 16.3 (30.0)

48. Secondary Outcome: Number of Participants With Biochemical Pregnancy, Clinical Pregnancy, Vital Pregnancy and Ongoing Pregnancy in Any of Treatment Cycles 1, 2 or 3
Description: Biochemical pregnancy: Pregnancy proven by a biochemical pregnancy test using urine samples or serum samples collected at least 14 days after ET. Participants not having a positive biochemical pregnancy test result, but with an ultrasound scan showing at least one gestational sac were counted as having a biochemical pregnancy. Clinical pregnancy: Presence of at least one gestational sac as assessed by ultrasound scan. Vital pregnancy: Presence of at least one fetus with heart activity as assessed by ultrasound scan. Ongoing pregnancy: Presence of at least one fetus with heart activity as assessed by ultrasound scan at least 10 weeks after ET, or confirmed by live birth.
Time Frame: ≥14 days (for biochemical pregnancy), 5-6 weeks (for clinical pregnancy), 5-6 weeks to 10 weeks (for vital pregnancy) and 10 weeks up to 9 months (for ongoing pregnancy) after ET, within a treatment cycle
Population: Participants who received corifollitropin alfa
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
participants
  Biochemical pregnancy | 340
  Clinical pregnancy | 303
  Vital pregnancy | 278
  Ongoing pregnancy | 272

49. Secondary Outcome: Number of Participants With Singleton and Multiple Ongoing Pregnancy in Any of Treatment Cycles 1, 2 or 3
Description: Singleton pregnancy is a pregnancy in which one fetus develops in the uterus. Multiple pregnancy is a pregnancy in which more than one fetus develops simultaneously in the uterus. Ongoing pregnancy: Presence of at least one fetus with heart activity as assessed by ultrasound scan at least 10 weeks after ET, or confirmed by live birth.
Time Frame: 10 weeks up to 9 months after ET, within a treatment cycle
Population: Participants who received corifollitropin alfa and had ongoing pregnancy in any of Treatment Cycles 1, 2 or 3
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 272
participants
  Singleton ongoing pregnancy | 226
  Multiple ongoing pregnancy | 46

50. Secondary Outcome: Number of Participants With Miscarriage Among Participants With Clinical Pregnancy in Any of Treatment Cycles 1, 2 or 3
Description: Miscarriage: Loss of the fetus without induction or instrumentation, also known as "spontaneous abortion." Clinical pregnancy: Presence of at least one gestational sac as assessed by ultrasound scan.
Time Frame: 5-6 weeks up to 9 months after ET, within a treatment cycle
Population: Participants who received corifollitropin alfa and had clinical pregnancy in any of Treatment Cycles 1, 2 or 3
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 303
participants | 37

51. Secondary Outcome: Number of Participants With Miscarriage Among Participants With Vital Pregnancy in Any of Treatment Cycles 1, 2 or 3
Description: Miscarriage: Loss of the fetus without induction or instrumentation, also known as "spontaneous abortion." Vital pregnancy: Presence of at least one fetus with heart activity as assessed by ultrasound scan.
Time Frame: 5-6 weeks up to 9 months after ET, within a treatment cycle
Population: Participants who received corifollitropin alfa and had vital pregnancy in any of Treatment Cycles 1, 2 or 3
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 278
participants | 5

52. Secondary Outcome: Number of Participants With Ectopic Pregnancy Among Participants With Biochemical Pregnancy in Any of Treatment Cycles 1, 2 or 3
Description: Ectopic pregnancy: A pregnancy in which the embryo attaches itself in a place other than inside the uterus. The most common site for an ectopic pregnancy is within one of the two fallopian tubes. Biochemical pregnancy: Pregnancy proven by a biochemical pregnancy test using urine samples or serum samples collected at least 14 days after ET. Participants not having a positive biochemical pregnancy test result, but with an ultrasound scan showing at least one gestational sac were counted as having a biochemical pregnancy.
Time Frame: From 2 weeks up to approximately 5-6 weeks after ET, within a treatment cycle
Population: Participants who received corifollitropin alfa and had biochemical pregnancy in any of Treatment Cycles 1, 2 or 3
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 340
participants | 9

53. Secondary Outcome: Number of Participants With Ongoing Pregnancy in Any FTET Cycle
Description: After the first and after the second treatment cycle (i.e., a cycle in which corifollitropin alfa was administered for ovarian stimulation), participants could continue with a maximum of three FTET cycles before starting the following treatment cycle. This measure summarizes the number of participants with ongoing pregnancy following ET within an FTET cycle. Ongoing pregnancy: Presence of at least one fetus with heart activity as assessed by ultrasound scan at least 10 weeks after ET, or confirmed by live birth.
Time Frame: 10 weeks up to 9 months after ET within an FTET cycle
Population: Participants who received corifollitropin alfa and had ET in any FTET cycle
Measure: Number; unit: participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 209
participants | 48

54. Secondary Outcome: Cumulative Ongoing Pregnancy Rate: Percentage of Participants With Ongoing Pregnancy in Treatment Cycles 1, 2 or 3, or in Any FTET Cycle, or Who Had Ongoing Pregnancy That Was a Spontaneous Pregnancy
Description: The ongoing pregnancy rate, cumulative over the entire study (in percent), is defined as 100 times the number of participants who had an ongoing pregnancy in Treatment Cycles 1, 2 or 3, or in any FTET cycle, or who had a spontaneous ongoing pregnancy, divided by the total number of participants who were administered corifollitropin alfa in the study. A participant could only be represented once in the count of ongoing pregnancies for determination of cumulative ongoing pregnancy rate. After the first and after the second treatment cycle (i.e., a cycle in which corifollitropin alfa was administered for ovarian stimulation), participants could continue with a maximum of three FTET cycles before starting the following treatment cycle. A spontaneous pregnancy is a pregnancy that was not considered to have resulted from ET in a treatment cycle or FTET cycle.
Time Frame: Up to approximately 26 months after first dose of corifollitropin alfa
Population: Participants who received corifollitropin alfa
Measure: Number; unit: percentage of participants
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 682
percentage of participants | 50.6

55. Secondary Outcome: Serum Follicle Stimulating Hormone (FSH) Levels in Treatment Cycle 1
Description: Blood samples for assessment of serum FSH were taken pre-dose (Stimulation Day 1), Stimulation Day 5 or 6 (prior to first GnRH antagonist administration), Stimulation Day 8, day of (rec)hCG administration, day of ET and 2 weeks after ET.
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: International Units (IU)/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 658
International Units (IU)/L
  Stimulation Day 1 (pre-dose) (n=651) | 7.18 (2.34)
  Stimulation Day 5 or 6 (n=648) | 24.00 (6.36)
  Stimulation Day 8 (n=634) | 13.23 (3.40)
  Day of (rec)hCG injection (n=643) | 13.63 (3.69)
  Day of embryo transfer (n=593) | 3.21 (1.68)
  2 weeks after embryo transfer (n=611) | 4.84 (3.51)

56. Secondary Outcome: Serum FSH Levels in Treatment Cycle 2
Description: as for outcome 55
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 364
IU/L
  Stimulation Day 1 (pre-dose) (n=357) | 7.17 (2.17)
  Stimulation Day 5 or 6 (n=358) | 24.24 (5.75)
  Stimulation Day 8 (n=346) | 13.38 (3.35)
  Day of (rec)hCG injection (n=358) | 13.78 (3.74)
  Day of embryo transfer (n=326) | 3.20 (1.45)
  2 weeks after embryo transfer (n=333) | 5.07 (3.33)

57. Secondary Outcome: Serum FSH Levels in Treatment Cycle 3
Description: as for outcome 55
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 190
IU/L
  Stimulation Day 1 (pre-dose) (n=185) | 7.50 (5.24)
  Stimulation Day 5 or 6 (n=186) | 24.51 (5.93)
  Stimulation Day 8 (n=184) | 13.56 (3.35)
  Day of (rec)hCG injection (n=183) | 13.62 (3.49)
  Day of embryo transfer (n=168) | 3.17 (1.55)
  2 weeks after embryo transfer (n=173) | 5.01 (3.40)

58. Secondary Outcome: Serum Luteinizing Hormone (LH) Levels in Treatment Cycle 1
Description: Blood samples for assessment of serum LH were taken pre-dose (Stimulation Day 1), Stimulation Day 5 or 6 (prior to first GnRH antagonist administration), Stimulation Day 8, day of (rec)hCG administration, day of ET and 2 weeks after ET.
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 658
IU/L
  Stimulation Day 1 (pre-dose) (n=651) | 5.07 (1.86)
  Stimulation Day 5 or 6 (n=648) | 4.86 (5.39)
  Stimulation Day 8 (n=634) | 1.34 (1.55)
  Day of (rec)hCG injection (n=643) | 1.53 (1.98)
  Day of embryo transfer (n=593) | NA (NA) — If more than 1/3 of the values per assessment day were smaller than the lower limit of quantitation (LLOQ) of the analytical method (0.6 IU/L), mean and SD are reported as missing.
  2 weeks after embryo transfer (n=611) | 3.27 (2.57)

59. Secondary Outcome: Serum LH Levels in Treatment Cycle 2
Description: as for outcome 58
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 364
IU/L
  Stimulation Day 1 (pre-dose) (n=357) | 5.13 (1.86)
  Stimulation Day 5 or 6 (n=358) | 4.78 (5.18)
  Stimulation Day 8 (n=346) | 1.35 (1.77)
  Day of (rec)hCG injection (n=358) | 1.67 (2.15)
  Day of embryo transfer (n=326) | NA (NA) — If more than 1/3 of the values per assessment day were smaller than the LLOQ of the analytical method (0.6 IU/L), mean and SD are reported as missing.
  2 weeks after embryo transfer (n=333) | 3.41 (2.48)

60. Secondary Outcome: Serum LH Levels in Treatment Cycle 3
Description: as for outcome 58
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 190
IU/L
  Stimulation Day 1 (pre-dose) (n=185) | 5.05 (1.97)
  Stimulation Day 5 or 6 (n=186) | 4.84 (5.39)
  Stimulation Day 8 (n=184) | 1.36 (1.50)
  Day of (rec)hCG injection (n=183) | 1.79 (2.71)
  Day of embryo transfer (n=168) | NA (NA) — If more than 1/3 of the values per assessment day were smaller than the LLOQ of the analytical method (0.6 IU/L), mean and SD are reported as missing.
  2 weeks after embryo transfer (n=173) | 3.57 (3.13)

61. Secondary Outcome: Serum Estradiol Levels in Treatment Cycle 1
Description: Blood samples for assessment of serum estradiol were taken pre-dose (Stimulation Day 1), Stimulation Day 5 or 6 (prior to first GnRH antagonist administration), Stimulation Day 8, day of (rec)hCG administration, day of ET and 2 weeks after ET.
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 658
pmol/L
  Stimulation Day 1 (pre-dose) (n=651) | 126.07 (74.36)
  Stimulation Day 5 or 6 (n=648) | 2246.72 (1479.01)
  Stimulation Day 8 (n=633) | 3224.72 (2013.62)
  Day of (rec)hCG injection (n=642) | 5602.90 (3400.47)
  Day of embryo transfer (n=593) | 2972.22 (1758.83)
  2 weeks after embryo transfer (n=611) | 1064.92 (2006.31)

62. Secondary Outcome: Serum Estradiol Levels in Treatment Cycle 2
Description: as for outcome 61
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 364
pmol/L
  Stimulation Day 1 (pre-dose) (n=357) | 120.80 (43.73)
  Stimulation Day 5 or 6 (n=357) | 2116.13 (1362.31)
  Stimulation Day 8 (n=346) | 3197.12 (2098.53)
  Day of (rec)hCG injection (n=358) | 5444.89 (2992.37)
  Day of embryo transfer (n=324) | 2988.11 (1823.81)
  2 weeks after embryo transfer (n=333) | 929.24 (1861.04)

63. Secondary Outcome: Serum Estradiol Levels in Treatment Cycle 3
Description: as for outcome 61
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 190
pmol/L
  Stimulation Day 1 (pre-dose) (n=185) | 117.5 (42.10)
  Stimulation Day 5 or 6 (n=185) | 1993.66 (1372.67)
  Stimulation Day 8 (n=184) | 3164.08 (2214.33)
  Day of (rec)hCG injection (n=183) | 5605.89 (3687.99)
  Day of embryo transfer (n=168) | 3065.47 (1988.36)
  2 weeks after embryo transfer (n=172) | 746.52 (1249.66)

64. Secondary Outcome: Serum Progesterone Levels in Treatment Cycle 1
Description: Blood samples for assessment of serum progesterone were taken pre-dose (Stimulation Day 1), Stimulation Day 5 or 6 (prior to first GnRH antagonist administration), Stimulation Day 8, day of (rec)hCG administration, day of ET and 2 weeks after ET.
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 658
nmol/L
  Stimulation Day 1 (pre-dose) (n=651) | 1.99 (2.40)
  Stimulation Day 5 or 6 (n=648) | 2.72 (11.85)
  Stimulation Day 8 (n=633) | 1.85 (2.00)
  Day of (rec)hCG injection (n=643) | 4.14 (23.37)
  Day of embryo transfer (n=593) | 331.16 (169.05)
  2 weeks after embryo transfer (n=611) | 100.31 (168.53)

65. Secondary Outcome: Serum Progesterone Levels in Treatment Cycle 2
Description: as for outcome 64
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 364
nmol/L
  Stimulation Day 1 (pre-dose) (n=357) | 1.84 (1.64)
  Stimulation Day 5 or 6 (n=358) | 2.14 (1.13)
  Stimulation Day 8 (n=346) | 1.75 (1.09)
  Day of (rec)hCG injection (n=358) | 3.91 (9.14)
  Day of embryo transfer (n=325) | 316.28 (174.25)
  2 weeks after embryo transfer (n=333) | 88.21 (165.39)

66. Secondary Outcome: Serum Progesterone Levels in Treatment Cycle 3
Description: as for outcome 64
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 190
nmol/L
  Stimulation Day 1 (pre-dose) (n=185) | 1.76 (0.74)
  Stimulation Day 5 or 6 (n=186) | 2.29 (3.37)
  Stimulation Day 8 (n=184) | 1.75 (0.74)
  Day of (rec)hCG injection (n=183) | 4.92 (14.81)
  Day of embryo transfer (n=168) | 311.64 (161.71)
  2 weeks after embryo transfer (n=173) | 79.03 (136.60)

67. Secondary Outcome: Serum Inhibin-B Levels in Treatment Cycle 1
Description: Blood samples for assessment of serum inhibin-B were taken pre-dose (Stimulation Day 1), Stimulation Day 5 or 6 (prior to first GnRH antagonist administration), Stimulation Day 8, day of (rec)hCG administration, day of ET and 2 weeks after ET.
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 1
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 658
pg/mL
  Stimulation Day 1 (pre-dose) (n=652) | 48.22 (29.91)
  Stimulation Day 5 or 6 (n=648) | 409.63 (299.19)
  Stimulation Day 8 (n=634) | 455.46 (372.09)
  Day of (rec)hCG injection (n=643) | 523.07 (464.36)
  Day of embryo transfer (n=591) | NA (NA) — If more than 1/3 of the values per assessment day were smaller than the LLOQ of the analytical method (10 pg/mL), mean and SD are reported as missing.
  2 weeks after embryo transfer (n=611) | NA (NA) — If more than 1/3 of the values per assessment day were smaller than the LLOQ of the analytical method (10 pg/mL), mean and SD are reported as missing.

68. Secondary Outcome: Serum Inhibin-B Levels in Treatment Cycle 2
Description: as for outcome 67
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 2
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 364
pg/mL
  Stimulation Day 1 (pre-dose) (n=356) | 48.88 (26.79)
  Stimulation Day 5 or 6 (n=358) | 406.29 (326.64)
  Stimulation Day 8 (n=346) | 443.32 (402.67)
  Day of (rec)hCG injection (n=358) | 505.02 (432.96)
  Day of embryo transfer (n=325) | 29.38 (34.99)
  2 weeks after embryo transfer (n=333) | 39.04 (33.74)

69. Secondary Outcome: Serum Inhibin-B Levels in Treatment Cycle 3
Description: as for outcome 67
Time Frame: Pre-dose (Stimulation Day 1) through 2 weeks after ET in Treatment Cycle 3
Population: Participants who received corifollitropin alfa and (rec)hCG injection in Treatment Cycle 3
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Corifollitropin Alfa 150 µg
Number analyzed (Participants) | 190
pg/mL
  Stimulation Day 1 (pre-dose) (n=185) | 50.49 (28.25)
  Stimulation Day 5 or 6 (n=186) | 406.14 (331.91)
  Stimulation Day 8 (n=184) | 439.83 (374.99)
  Day of (rec)hCG injection (n=183) | 504.03 (437.68)
  Day of embryo transfer (n=168) | 26.28 (25.03)
  2 weeks after embryo transfer (n=173) | 40.16 (34.05)

ADVERSE EVENTS:
Time Frame: Up to approximately 26 months after first dose of corifollitropin alfa
Description: SAEs that occurred in fetuses or infants during the study period are included in the summary of SAEs, and are allocated to the associated study participant who was administered corifollitropin alfa.
Arm/Group | Corifollitropin Alfa 150 µg
Serious Adverse Events (participants affected / at risk) | 51/682
Other Adverse Events (participants affected / at risk) | 239/682
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 150 µg (N=682)
Autosomal chromosome anomaly (Congenital, familial and genetic disorders) | 1 (2)
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1 (1)
Congenital uterine anomaly (Congenital, familial and genetic disorders) | 1 (1)
Cytogenetic abnormality (Congenital, familial and genetic disorders) | 1 (1)
Ectopia cordis (Congenital, familial and genetic disorders) | 1 (1)
Encephalocele (Congenital, familial and genetic disorders) | 1 (1)
Trisomy 15 (Congenital, familial and genetic disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Growth retardation (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 3 (3)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Arrested labour (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Heterotopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Placenta praevia haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 3 (5)
Premature labour (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Retroplacental haematoma (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Small for dates baby (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Twin pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Psychosomatic disease (Psychiatric disorders) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 2 (2)
Fallopian tube disorder (Reproductive system and breast disorders) | 1 (1)
Ovarian haematoma (Reproductive system and breast disorders) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 10 (10)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Uterine cervix stenosis (Reproductive system and breast disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric stapling reversal (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Corifollitropin Alfa 150 µg (N=682)
Procedural pain (Injury, poisoning and procedural complications) | 121 (163)
Headache (Nervous system disorders) | 62 (91)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 48 (51)
Pelvic discomfort (Reproductive system and breast disorders) | 35 (39)
Pelvic pain (Reproductive system and breast disorders) | 51 (60)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publications must be based on data validated and released by the Sponsor. Any scientific paper, presentation, or other communication concerning the study must first be submitted to the Sponsor, at least 6 weeks prior to estimated publication or presentation, for written consent. Sponsor has the right to make its consent conditional upon proper representation of the interpretation of both the Sponsor and the Investigator in the discussion of the data in such communications.